CLINICAL TRIAL: NCT04341025
Title: Providing Insight Into and Mindfulness for Situational Erectile Dysfunction
Acronym: PRIMED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vancouver Coastal Health (Other Government)
Responsible Party: Principal Investigator, Miriam Driscoll, PI, Vancouver Coastal Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H18-00665
Record Dates: First submitted 2019-06-27; First posted 2020-04-10 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Situational Erectile Dysfunction
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Participants will take part in a 6-session MBPST group for treatment of situational ED. Each session will be 2 hours in length and will be spaced one week apart, for a total of 12 hours of treatment time. Participants will also take part in supportive group follow-up sessions at 1- and 4-months following group completion. Treatment endpoints will be assessed at four time-points (pre-treatment, immediate post-treatment, 1-month post-treatment, and 4-months post-treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Patients are compared to themselves before and after the treatment.
  Interventions: Behavioral: Mindfulness based psychosexual therapy ( MBPST)

INTERVENTIONS:
Behavioral: Mindfulness based psychosexual therapy ( MBPST) — The group treatment sessions will integrate empirically supported elements of psychoeduation, cognitive behavioural therapy, and mindfulness skills. Each of the six sessions will follow the well-defined manualized treatment protocol. The treatment is adapted from the study team's previous mindfulness-based treatment group (H15-03172), for situational ED which has been shown to be effective. Participants will be provided with handouts and asked to complete approximately 10-60 minutes/day of at-home practice/skills, which may include reading material, mindfulness exercises, and/or behavioural exercises between sessions. During the 2 follow-up sessions, participants will be invited to share their experience since the conclusion of group, ask questions, and participate in troubleshooting.
  Other Names: MBCT ( Mindfulness based cognitive therapy )

SUMMARY:
Erectile dysfunction (ED) is among the most common sexual dysfunctions experienced by men, affecting at least one third of men across the lifespan. Although pharmacological treatments are available, adherence to these treatments is poor, suggesting the need for integration of psychological interventions. This study will determine if a 6-session mindfulness-based psychosexual therapy (MBPST) group will be effective and feasible for men with situational ED. This study is adapted from a previously published 4-session MBPST protocol which was found to be beneficial for men with situational ED. Outcomes are measured using self-report questionnaires on sexual functioning/enjoyment, relationship satisfaction, and treatment acceptability.

DETAILED DESCRIPTION:
PURPOSE The purpose of this study is to assess the feasibility and efficacy of a 6-session mindfulness-based psychosexual therapy (MBPST) treatment protocol using self-report questionnaires. The current protocol is adapted from a pre-existing 4-session mindfulness-based psychosexual therapy (MBPST) protocol from a pilot study which has already demonstrated benefits in the treatment of situational erectile dysfunction (ED). The six sessions include elements of psychoeducation, cognitive therapy, mindfulness training, and sex therapy techniques. The elements comprising the six sessions are evidence-based, as their effectiveness has been demonstrated in female samples (e.g., Brotto et al., 2012; Paterson et al., 2017), and more recently in the context of a four-session pilot in men with situational ED (H15-03172; published in Bossio et al., 2018). The rationale for an increase from a 4 to 6-session approach came from qualitative analysis of participant perspectives in the pilot study and from investigator experience.

HYPOTHESES

1. Men who undergo MBPST treatment will show significant post-treatment improvements at follow-up (immediately following treatment and at 1- and 4-months after treatment completion), compared to baseline, to primary endpoints of: (i) erectile functioning; (ii) sexual distress; (iii) sexual satisfaction and pleasure.
2. Men who undergo MBPST treatment will show significant post-treatment improvements at follow-up (immediately following treatment and at 1- and 4-months after treatment completion), compared to baseline, to secondary endpoints of: (i) psychological variables/mental status (i.e., anxiety); (ii) mindfulness-related variables; and (iii) relationship satisfaction. The role of secondary endpoints as mediators to primary endpoints of sexual functioning will also be assessed.
3. Men will report significantly less use of medications for ED (i.e., PDE5 inhibitors and intracavernosal injections) at 4-month follow-up compared to pre-treatment.

JUSTIFICATION Sexual dysfunction affects at least one third of men across the lifespan (Laumann, Paik, & Rosen, 1999), and can have significant impact on quality of life and on intimate relationships (Hatzimouratidis et al., 2010). Erectile dysfunction (ED), or the inability to attain and/or maintain an erection sufficient for satisfactory sexual activity (NIH, 1993), is among the most common sexual dysfunctions experienced by men. The aetiology of ED is complex and can result from a variety of physiological (e.g., age, cardiovascular health, medication use), psychological (e.g., anxiety), and lifestyle factors (e.g., smoking status; Nicolosi, Moreira, Shirai, Tambi, & Glasser, 2003). Situational ED refers to ED that occurs in certain contexts (e.g., with a partner), but not others (e.g., masturbation, nocturnal erections).

Although pharmacological interventions (i.e., PDE5 inhibitors) have been available to treat ED since the 1990's, adherence to these treatments is poor, with approximately 50% of men failing to re-fill their first prescription (Carvalheira, Pereira, Maroco, & Forjaz, 2012; Hanash, 1997), despite the restoration of erections (Giannitsas, Konstantinopoulos, Patsialas, & Perimenis, 2008). This low adherence to pharmacological treatments suggests that there are aspects of ED, beyond the rigidity of erections that are not being addressed by medications. This may be particularly true in the case of situational ED, where psychogenic factors are playing a major role (McCabe et al., 2016).

There is increasing evidence documenting the benefits of MBCT for women with sexual dysfunction (Brotto, Basson, & Luria, 2008; Brotto et al., 2008; Brotto et al., 2012; Brotto, Seal, & Rellini, 2012; Brotto & Basson, 2014; Paterson, Handy, & Brotto, 2017). Further, the investigators recently adapted a pre-existing 4-session MBPST protocol, which had already been shown to be effective in the treatment of female sexual dysfunction, to fit the needs of men with situational ED and pilot-tested it in group format (H15-03172). Our pilot data suggest significant benefits for men with situational ED (Bossio, Basson, Driscoll, Correia, & Brotto, 2019). However, feedback from the pilot participants indicated a need for additional sessions as they had only begun to establish a regular mindfulness practice. Mindfulness-based interventions consisting of eight sessions are common and have been shown to be effective in reducing depressive symptoms (Sipe & Eisendrath, 2012), depressive relapse (Teasdale, Segal, Williams, Ridgeway, Soulsby, & Lau, 2000), and anxiety (Evans, Ferrando, Findler, Stowell, Smart, & Haglin, 2008). However, the investigators were skeptical about the willingness and ability of patients to commit to eight consecutive weeks of treatment. Therefore, the current project is a pilot study intended to assess the feasibility and efficacy of a 6-session MBPST program for situational ED.

OBJECTIVES The main objective of this study is to test the feasibility and efficacy of a 6-session MBPST protocol for men with situational ED. Specifically, the investigators hope to find that men who undergo this treatment will experience improvements in primary (e.g., decreased erectile dysfunction and sexual distress), and secondary endpoints (e.g., increased relationship satisfaction and mental well-being). Further, the investigators hope to find that gains in the primary and secondary endpoints are maintained at 1- and 4-months.

RESEARCH DESIGN Participants (N=60) will take part in a 6-session MBPST group (n=6-10) for treatment of situational ED, either in-person or in an online format. Each session will be 2 hours in length and will be spaced one week apart, for a total of 12 hours of treatment time. Participants will also take part in supportive group follow-up sessions at 1- and 4-months following group completion where participants are free to share their experiences with the group, ask questions, and participate in troubleshooting. Treatment endpoints will be assessed at four time-points (pre-treatment (Time 1), immediate post-treatment (Time 2), 1-month post-treatment (Time 3), and 4-months post-treatment (Time 4)).

STATISTICAL ANALYSIS One-way repeated-measures multivariate analysis of variance (MANOVA) will be used to assess our primary hypothesis-that men will show improvements in primary (i.e., sexual functioning) endpoints following treatment-with the primary endpoint measures as the dependent variables (e.g., ED severity, sexual distress, sexual satisfaction, pleasure), time-point (pre-treatment, immediate post-treatment, 1-month post-treatment, and 4-months post-treatment) as the independent variable, and age as a covariate.

Our secondary hypotheses-that men will show improvements secondary endpoints (i.e., mindfulness-related variables, mental status, and relationship factors) following treatment-will also be examined using the same repeated-measures MANOVA strategy described above. The hypothesis that secondary endpoints act as mediators of sexual functioning following treatment will also be examined using repeated-measures ANOVAs with primary endpoint measures as the dependent variable (i.e., sexual functioning), time-point (pre-treatment, immediate post-treatment, 1-month post-treatment, and 4-months post-treatment) as the independent variable, and secondary endpoints (e.g., change in relationship satisfaction) as mediators.

Our tertiary hypothesis-that men will report using medications for ED significantly less 4-months after treatment conclusion compared with pre-treatment use-will be assessed using paired-sample t-tests comparing frequency of use and dose before treatment and 4-months after treatment.

ELIGIBILITY:
Inclusion Criteria:

This study is open to individuals who are:

* Diagnosed with situational erectile dysfunction (ED) of at least 6 months duration, as assessed by a physician at the BC Centre for Sexual Medicine according to DSM-5 criteria
* 19 years of age or older
* Fluent enough in English to participate in group
* Willing to abstain from using medications for ED (i.e., PDE5 inhibitors, intracavernosal injections, MUSE etc.) from the start of treatment until the 1-month follow-up (totaling 10 weeks)
* Comfortable and interested in participating in a small group format with 6-10 others

Exclusion Criteria:

This study is not suitable for individuals who:

* Do not experience an exacerbation of ED in the partnered context
* Have a current unmanaged health condition (e.g., unmanaged diabetes mellitus) or unstable mental health condition (e.g., severe depression/anxiety, active suicidal ideation) that would interfere with self- or partnered-sexual activities or with group participation
* Do no feel comfortable participating in a small group format with 6-10 others

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported Erectile Functioning as measured by International Index of Erectile Function - 5 | Change from baseline to immediately post treatment (6 weeks)
  (IIEF-5; Rosen, Cappelleri, Smith, Lipsky, & Pena, 1999); 5 item questionnaire
Self-reported Erectile Functioning as measured by International Index of Erectile Function - 5 | Change from baseline to one month post-treatment (10 weeks)
  (IIEF-5; Rosen, Cappelleri, Smith, Lipsky, & Pena, 1999); 5 item questionnaire
Self-reported Erectile Functioning as measured by International Index of Erectile Function - 5 | Change from baseline to four months post-treatment (22 weeks)
  (IIEF-5; Rosen, Cappelleri, Smith, Lipsky, & Pena, 1999); 5 item questionnaire
Self-reported Sexual Distress as measured by Sexual Distress Scale-Revised | Change from baseline to immediately post treatment (6 weeks)
  (Derogatis, Clayton, Lewis-D'Agostino, Wunderlich, & Fu, 2008). This scale was recently validated for measuring sexual distress in men (Santos-Iglesias, Mohamed, Danko, & Walker, 2018); 13 item rating scale
Self-reported Sexual Distress as measured by Sexual Distress Scale-Revised | Change from baseline to one month post-treatment (10 weeks)
  (Derogatis, Clayton, Lewis-D'Agostino, Wunderlich, & Fu, 2008). This scale was recently validated for measuring sexual distress in men (Santos-Iglesias, Mohamed, Danko, & Walker, 2018); 13 item rating scale
Self-reported Sexual Distress as measured by Sexual Distress Scale-Revised | Change from baseline to four months post-treatment (22 weeks)
  (Derogatis, Clayton, Lewis-D'Agostino, Wunderlich, & Fu, 2008). This scale was recently validated for measuring sexual distress in men (Santos-Iglesias, Mohamed, Danko, & Walker, 2018); 13 item rating scale
Self-reported Confidence in Sexual and Erectile Competence as measured by Sexual Self-Efficacy Scale - Erectile Functioning | Change from baseline to immediately post treatment (6 weeks)
  (Fichten, Spector, Amsel, Creti, Brender, & Libman, 1998), which measures confidence in sexual and erectile competence; 25 item rating scale
Self-reported Confidence in Sexual and Erectile Competence as measured by Sexual Self-Efficacy Scale - Erectile Functioning | Change from baseline to one month post-treatment (10 weeks)
  (Fichten, Spector, Amsel, Creti, Brender, & Libman, 1998), which measures confidence in sexual and erectile competence; 25 item rating scale
Self-reported Confidence in Sexual and Erectile Competence as measured by Sexual Self-Efficacy Scale - Erectile Functioning | Change from baseline to four months post-treatment (22 weeks)
  (Fichten, Spector, Amsel, Creti, Brender, & Libman, 1998), which measures confidence in sexual and erectile competence; 25 item rating scale
Self-reported Sexual Satisfaction and Pleasure as measured by International Index of Erectile Function - Overall Satisfaction Subscale. | Change from baseline to immediately post treatment (6 weeks)
  (Rosen, Riley, Wagner, Osterloh, Kirkpatrick, & Mishra, 1997), which measures sexual satisfaction. 2-item questionnaire
Self-reported Sexual Satisfaction and Pleasure as measured by International Index of Erectile Function - Overall Satisfaction Subscale | Change from baseline to one month post-treatment (10 weeks)
  (Rosen, Riley, Wagner, Osterloh, Kirkpatrick, & Mishra, 1997), which measures sexual satisfaction. 2-item questionnaire
Self-reported Sexual Satisfaction and Pleasure as measured by International Index of Erectile Function - Overall Satisfaction Subscale | Change from baseline to four months post-treatment (22 weeks)
  (Rosen, Riley, Wagner, Osterloh, Kirkpatrick, & Mishra, 1997), which measures sexual satisfaction. 2-item questionnaire
Self-reported Sexual Pleasure as measured by an investigator-created Questionnaire | Change from baseline to immediately post treatment (6 weeks)
  2-item self report questionnaire on a 5-point scale assessing physical and emotional sexual pleasure.
Self-reported Sexual Pleasure as measured by an investigator-created Questionnaire | Change from baseline to one month post-treatment (10 weeks)
  2-item self report questionnaire on a 5-point scale assessing physical and emotional sexual pleasure.
Self-reported Sexual Pleasure as measured by an investigator-created Questionnaire | Change from baseline to four months post-treatment (22 weeks)
  2-item self report questionnaire on a 5-point scale assessing physical and emotional sexual pleasure.

SECONDARY OUTCOMES:
Anxiety Symptoms as measured by Generalized Anxiety Disorder-7 | Change from baseline to immediately post treatment (6 weeks)
  (Spitzer, Kroenke, Williams, & Lowe, 2006),7-item questionnaire
Anxiety Symptoms as measured by Generalized Anxiety Disorder-7 | Change from baseline to one month post-treatment (10 weeks)
  (Spitzer, Kroenke, Williams, & Lowe, 2006), 7-item questionnaire
Anxiety Symptoms as measured by Generalized Anxiety Disorder-7 | Change from baseline to four months post-treatment (22 weeks)
  (Spitzer, Kroenke, Williams, & Lowe, 2006), 7-item questionnaire
Degree of Mindfulness as measured by the Five Facet Mindfulness Questionnaire-15 | Change from baseline to immediately post treatment (6 weeks)
  (Baer, Carmody, Hunsinger, 2012; Gu, Strauss, Crane, Barnhofer, Karl, Cavanagh, & Kuyken, 2016),15-item questionnaire
Degree of Mindfulness as measured by the Five Facet Mindfulness Questionnaire-15 | Change from baseline to one month post-treatment (10 weeks)
  (Baer, Carmody, Hunsinger, 2012; Gu, Strauss, Crane, Barnhofer, Karl, Cavanagh, & Kuyken, 2016),15-item questionnaire
Degree of Mindfulness as measured by the Five Facet Mindfulness Questionnaire-15 | Change from baseline to four months post-treatment (22 weeks)
  (Baer, Carmody, Hunsinger, 2012; Gu, Strauss, Crane, Barnhofer, Karl, Cavanagh, & Kuyken, 2016),15-item questionnaire
Non-attachment mindfulness skill as measured by Nonattachment Scale-7 | Change from baseline to immediately post treatment (6 weeks)
  (Sahdra, Ciarrochi, Parker, Marshall, & Heaven, 2015) Non-attachment is a specific facet of mindfulness measured by this 7-item questionnaire
Non-attachment mindfulness skill as measured by Nonattachment Scale-7 | Change from baseline to one month post-treatment (10 weeks)
  (Sahdra, Ciarrochi, Parker, Marshall, & Heaven, 2015) Non-attachment is a specific facet of mindfulness measured by this 7-item questionnaire
Non-attachment mindfulness skill as measured by Nonattachment Scale-7 | Change from baseline to four months post-treatment (22 weeks)
  (Sahdra, Ciarrochi, Parker, Marshall, & Heaven, 2015) Non-attachment is a specific facet of mindfulness measured by this 7-item questionnaire
Relationship satisfaction as measured by Relationship Assessment Scale | Change from baseline to immediately post treatment (6 weeks)
  (Hendrick, 1988) 7-item questionnaire
Relationship satisfaction as measured by Relationship Assessment Scale | Change from baseline to one month post-treatment (10 weeks)
  (Hendrick, 1988) 7-item questionnaire
Relationship satisfaction as measured by Relationship Assessment Scale | Change from baseline to four months post-treatment (22 weeks)
  (Hendrick, 1988)7-item questionnaire

OTHER OUTCOMES:
Patient Satisfaction towards therapy group and Self-reported Impact on Quality of Sexual Life as measured by Patient Global Impression of Change Scale - Revised | Change from baseline to immediately post treatment (6 weeks)
  (adapted from Hurst & Bolton, 2004) This is a single self-report question on participants overall satisfaction from and impact from the treatment group
Patient Satisfaction towards therapy group and Self-reported Impact on Quality of Sexual Life as measured by Patient Global Impression of Change Scale - Revised | Change from baseline to one month post-treatment (10 weeks)
  (adapted from Hurst & Bolton, 2004). This is a single self-report question on participants overall satisfaction from and impact from the treatment group
Patient Satisfaction towards therapy group and Self-reported Impact on Quality of Sexual Life as measured by Patient Global Impression of Change Scale - Revised | Change from baseline to four months post-treatment (22 weeks)
  (adapted from Hurst & Bolton, 2004) This is a single self-report question on participants overall satisfaction from and impact from the treatment group
PDE5 inhibitor Medication Use | Change from baseline to immediately post treatment (6 weeks)
  As measured by self-report questions asking men about their use of PDE5 inhibitor medications to erectile functioning, and their perception of these medications usefulness
PDE5 inhibitor Medication Use | Change from baseline to one month post-treatment (10 weeks)
  As measured by self-report questions asking men about their use of PDE5 inhibitor medications to erectile functioning, and their perception of these medications usefulness
PDE5 inhibitor Medication Use | Change from baseline to four months post-treatment (22 weeks)
  As measured by self-report questions asking men about their use of PDE5 inhibitor medications to erectile functioning, and their perception of these medications usefulness
Mindfulness and Sexual Activities Practice as measured by investigator-created questionnaire | Change from baseline to immediately post treatment (6 weeks)
  Daily log of types of activities and minutes practiced
Mindfulness and Sexual Activities Practice as measured by investigator-created questionnaire | Change from baseline to one month post-treatment (10 weeks)
  Daily log of types of activities and minutes practiced
Mindfulness and Sexual Activities Practice as measured by investigator-created questionnaire | Change from baseline to four months post-treatment (22 weeks)
  Daily log of types of activities and minutes practiced

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Driscoll, MD, Principal Investigator — UBC
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bossio JA, Basson R, Driscoll M, Correia S, Brotto LA. Mindfulness-Based Group Therapy for Men With Situational Erectile Dysfunction: A Mixed-Methods Feasibility Analysis and Pilot Study. J Sex Med. 2018 Oct;15(10):1478-1490. doi: 10.1016/j.jsxm.2018.08.013. PMID 30297094